CLINICAL TRIAL: NCT06386757
Title: Comparison Between Nasal and Oropharyngeal Bleeding in Video Laryngoscopy and Direct Laryngoscopy for Nasal Intubation in Maxillofacial Trauma Patients: a Randomized Controlled Trial
Brief Title: Comparison Between Nasal and Oropharyngeal Bleeding in Video Laryngoscopy and Direct Laryngoscopy for Nasal Intubation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Soudy Salah Hammad, Lecturer of anesthesia and surgical intensive care, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Asw.U. 911/3/24
Record Dates: First submitted 2024-04-04; First posted 2024-04-26 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Maxillofacial Injuries; Nasal Bleeding; Intubation Complication
Keywords: nasal intubation; videolaryngscopy; direct laryngscopy; bogie stylet
MeSH Terms: conditions — Maxillofacial Injuries; Epistaxis

STUDY DESIGN:
Intervention Model Description: These prospective, randomized, controlled clinical trials will be conducted at Aswan University Hospital on 62 patients who are scheduled for maxillofacial surgeries requiring nasal intubation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Ι Combined Video Laryngoscopy (VL) and Bougie (Active Comparator): Group Ι Combined Video Laryngoscopy (VL) and Bougie: Nasal intubation will be performed using a video laryngoscope and a bougie.
- Group ΙI Direct Laryngoscopy (DL) and Bougie : (Active Comparator): Nasal intubation will be performed using a traditional direct laryngoscope and a bougie.
  Interventions: Procedure: Combined Direct Laryngoscopy (DL) and Bougie

INTERVENTIONS:
Procedure: Combined Video Laryngoscopy (VL) and Bougie — To compare combined video laryngoscopy and bougie versus direct laryngoscopy and bougie for nasal intubation.
Procedure: Combined Direct Laryngoscopy (DL) and Bougie — To compare combined video laryngoscopy and bougie versus direct laryngoscopy and bougie for nasal intubation
  Arms: Group ΙI Direct Laryngoscopy (DL) and Bougie :

SUMMARY:
The objective of this study is to compare the effectiveness and safety of video laryngoscopy versus direct laryngoscopy for nasal intubation in patients with maxillofacial fractures regarding less bleeding to oral and nasal structures, quicker intubation times, increased success rates for first intubation attempts, fewer uses of the Magill forceps and the less need for cervical spine extension

DETAILED DESCRIPTION:
Maxillofacial fractures occur in a significant proportion worldwide and can occur as an isolated injury or in combination with other severe injuries including cranial, spinal, and upper and lower body injuries requiring prompt diagnosis with possible emergency interventions. The epidemiology of facial fractures varies with regard to injury type, severity, and cause and depends on the population studied.

Traumatic maxillofacial fractures are known to have difficulty in airway management due to anatomical and functional reasons. In many situations, treatment of facial fractures requires tracheal intubation. For fractures that involve occlusion, such as mandibular and Lefort fractures, oral intubation inhibits appropriate resolution of the occlusion. In these situations, nasotracheal intubation is indicated.

Direct laryngoscopic (DL) nasal intubations may be challenging if there is altered airway anatomy, difficulty in advancing the endotracheal tube through the glottis or in providers who are in training or those with less experience, even for patients with normal airway anatomy. The presence of cervical spine injury limit neck extension and makes airway manipulation more difficult. The use of Magill forceps is not always successful and is associated with endotracheal tube cuff damage and postoperative pharyngitis.

Video laryngoscopy (VL) is an adjunctive technique in anesthesia that utilizes a camera at the tip of the laryngoscope blade, which provides an indirect view of the glottis and surrounding structures during intubation displayed on a monitor. Use of video laryngoscopes has been shown to result in higher first intubation success, better laryngoscopic views, less mucosal trauma.

A bougie that is a long, stiff plastic wand is required to direct the tube to the glottis through manipulation through nasal route. bougie overcame the limitations of endotracheal tube direction and provided an advantage of rail-roading the tube over the bougie under vision leaving no possibility of trauma caused by direct or magill forceps tube manipulation.

Epistaxis is the most common complication encountered during nasotracheal (NT) intubation and may have serious consequences, such as lifethreatening bleeding and airway obstruction by aspirated blood. In addition, it may occur even when mucosal vasoconstriction, a lubricated tracheal tube and careful manipulation of the tube during insertion are employed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo maxillofacial surgeries with nasotracheal intubation..
* ASA I/II patients.
* BMI <35

Exclusion Criteria:

* Having bleeding diathesis and abnormal Prothrombin Time (PT), Partial Thromboplastin Time (PTT), or platelet counts.
* Local causes of bleeding as adenoid
* On medications that alter blood coagulation as anticoagulants and antiplatlets.
* Patients in which either intubation failed on both nostrils or where intubation was only possible with a tube smaller than 6.0 mm internal diameter(ID).
* Anticipated difficult airways.
* ASA III/IV.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of nasal and oropharyngeal bleeding | Through study completion, average 60 minutes at 5, 15, 30 minutes
  Incidence of nasal and oropharyngeal bleeding using Fromme's ordinal scale which is used for assessment of the surgical field quality( V Rajanigandha, et al. 2023),we will modify this scale to evaluate airway as follows :
  0- No bleeding (virtually bloodless field)
  1. Minimal bleeding ( not a nuisance to vision , no suctioning required)
  2. Mild bleeding (a nuisance to vision but does not compromises laryngeal tube insertion, occasional suctioning required )
  3. Moderate bleeding (slightly compromises laryngeal tube insertion, frequent suctioning required)
  4. Severe bleeding (significantly compromises laryngeal tube insertion, frequent suctioning required)
  5. Massive bleeding (cannot insert laryngeal tube, constant suctioning required)

SECONDARY OUTCOMES:
Time of successful intubation, defined as the time from removal of mask ventilation and beginning of bougie insertion until inflation of tube cuff | Within minutes
  Time of successful intubation, defined as the time from removal of mask ventilation and beginning of bougie insertion until inflation of tube cuff
Overall rate of first trial success. | Within minutes
  Overall rate of first trial success.
The use of magill forceps | Within minutes
  The use of magill forceps

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Alazhary, MD, Principal Investigator — Aswan University; Ayman M Eldemrdash, MD, Principal Investigator — Aswan University
Locations (1):
- Aswan University, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nedrud SM, Baasch DG, Cabral JD, McEwen DS, Dasika J. Combined Video Laryngoscope and Fiberoptic Nasal Intubation. Cureus. 2021 Nov 11;13(11):e19482. doi: 10.7759/cureus.19482. eCollection 2021 Nov. PMID 34912623
- [Background] Kumar P, Sharma J, Johar S, Singh V. Guiding Flexible-Tipped Bougie Under Videolaryngoscopy: An Alternative to Fiberoptic Nasotracheal Intubation in Maxillofacial Surgeries. J Maxillofac Oral Surg. 2020 Jun;19(2):324-326. doi: 10.1007/s12663-020-01327-w. Epub 2020 Jan 24. PMID 32346248
- [Background] Prasant MC, Kar S, Rastogi S, Hada P, Ali FM, Mudhol A. Comparative Study of Blood Loss, Quality of Surgical Field and Duration of Surgery in Maxillofacial Cases with and without Hypotensive Anesthesia. J Int Oral Health. 2014 Nov-Dec;6(6):18-21. PMID 25628477
- [Derived] Eldemrdash AM, Alazhary MA, Zaher ZZ, Hemaida TS, Yahia ME, Hammad SS. Comparison of Nasal and Oropharyngeal Bleeding in Video Laryngoscopy Versus Direct Laryngoscopy for Nasotracheal Intubation in Maxillofacial Trauma: A Randomized Controlled Trial. Anesthesiol Res Pract. 2025 Jul 3;2025:7797828. doi: 10.1155/anrp/7797828. eCollection 2025. PMID 40642178